CLINICAL TRIAL: NCT04239092
Title: Phase 1 Study of 9-ING-41, a Glycogen Synthase Kinase 3 Beta (GSK 3β) Inhibitor, as a Single Agent or With Irinotecan, Irinotecan Plus Temozolomide, or With Cyclophosphamide Plus Topotecan in Pediatric Patients With Refractory Malignancies.
Brief Title: 9-ING-41 in Pediatric Patients With Refractory Malignancies.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The decision to conclude study was made to optimize the clinical study design and protocol to further evaluate the safety profile of elraglusib (9-ING-41) in pediatric and adult patients with refractory Ewings Sarcoma.
Sponsor: Actuate Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1902
Record Dates: First submitted 2020-01-20; First posted 2020-01-23 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Refractory Cancer; Refractory Neoplasm; Cancer Pediatric; Refractory Tumor; Pediatric Cancer; Pediatric Brain Tumor; Neuroblastoma; Neuroblastoma Recurrent; Pediatric Lymphoma; Pediatric Meningioma; Diffuse Intrinsic Pontine Glioma
Keywords: 9-ING-41; GSK3beta; Glycogen Synthase Kinase 3 Beta inhibitor; ATR/Chk1
MeSH Terms: conditions — Neoplasms; Neuroblastoma; Meningioma; Diffuse Intrinsic Pontine Glioma | interventions — 3-(5-fluorobenzofuran-3-yl)-4-(5-methyl-5H-(1,3)dioxolo(4,5-f)indol-7-yl)-pyrrole-2,5-dione; Irinotecan; Temozolomide; Cyclophosphamide; Topotecan

STUDY DESIGN:
Intervention Model Description: Patients will received either single agent 9-ING-41 or 9-ING-41 plus Irinotecan or 9-ING-41 plus Irinotecan plus Temozolomide or 9-ING-41 plus Cyclophosphamide plus Topotecan
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 9-ING-41 (Experimental): 9-ING-41 will be administered by intravenous infusion twice weekly at an initial dose of 9.3 mg/kg. Cycle duration is 21 days.
  Interventions: Drug: 9-ING-41
- 9-ING-41 plus Irinotecan (Experimental): 9-ING-41 will be administered by intravenous infusion twice weekly at an initial dose of 9.3 mg/kg. Irinotecan will be administered at a dose of 50 mg/m2/day over 90 minutes IV on days 1-5 every 21 days (cycle duration is 21 days).
  Interventions: Drug: 9-ING-41; Drug: Irinotecan
- 9-ING-41 plus Irinotecan plus Temozolomide (Experimental): 9-ING-41 will be administered by intravenous infusion twice weekly at an initial dose of 9.3 mg/kg. Irinotecan will be administered at a dose of 50 mg/m2/day over 90 minutes IV on days 1-5 every 21 days. Temozolomide will be administered at a dose of 100 mg/m2/dose by mouth on Days 1 through 5 ((cycle duration is 21 days).
  Interventions: Drug: 9-ING-41; Drug: Irinotecan; Drug: Temozolomide
- 9-ING-41 plus Cyclophosphamide plus Topotecan (Experimental): Cyclophosphamide 400 mg/m2/dose administered intravenously over 30 min on Days 1 through 5. Topotecan 1.2 mg/m2/dose administered intravenously over 30 min once on Days 1 through 5. 9-ING-41 intravenous infusion twice weekly (cycle duration is 21 days).
  Interventions: Drug: 9-ING-41; Drug: Cyclophosphamide; Drug: Topotecan

INTERVENTIONS:
Drug: 9-ING-41 — 9-ING-41 will be administered by intravenous infusion twice weekly at an initial dose of 9.3 mg/kg. Cycle duration is 21 days.
  Other Names: 9-ING-41 COMPOUND
Drug: Irinotecan — Irinotecan 50 mg/m2/day administered over 90 minutes IV on days 1-5 every 21 days.
  Other Names: CPT-11
  Arms: 9-ING-41 plus Irinotecan; 9-ING-41 plus Irinotecan plus Temozolomide
Drug: Temozolomide — Temozolomide will be administered at a dose of 100 mg/m2/dose by mouth on Days 1 through 5 of a 21 day cycle.
  Other Names: Temodar
  Arms: 9-ING-41 plus Irinotecan plus Temozolomide
Drug: Cyclophosphamide — Cyclophosphamide 400 mg/m2/dose administered intravenously over 30 min on Days 1 through 5 of a 21 day cycle.
  Other Names: Cyclophosphamide IV
  Arms: 9-ING-41 plus Cyclophosphamide plus Topotecan
Drug: Topotecan — Topotecan 1.2 mg/m2/dose administered intravenously over 30 min once on Days 1 through 5 of a 21 day cycle.
  Other Names: Topotecan IV
  Arms: 9-ING-41 plus Cyclophosphamide plus Topotecan

SUMMARY:
9-ING-41 has anti-cancer clinical activity with no significant toxicity in adult patients. This Phase 1 study will study its efficacy in paediatric patients with advanced malignancies.

DETAILED DESCRIPTION:
9-ING-41 is a first-in-class, intravenously administered, maleimide-based, small molecule, potent selective GSK-3β inhibitor with significant pre-clinical and clinical anticancer activity. In the ongoing Actuate 1801 study in a cohort of over 90 patients with advanced refractory malignancies, 9-ING-41 has exhibited no significant toxicity, including no myelosuppression, and significant anti-tumor activity. 9-ING-41 also has significant pre-clinical ability to reverse pathologic fibrosis in multiple models of pulmonary and pleural fibrosis. 9-ING-41 is very highly active against neuroblastoma in diverse pre-clinical models. This Phase 1 study is designed to evaluate the safety and efficacy of 9-ING-41, as a single agent or in combination with irinitecan, in paediatric patients with advanced malignancies and thus to establish the recommended Phase 2 dose (RP2D) for further paediatric patient studies.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet ALL the following criteria to be eligible for this study:

1. Age < 22 years of age
2. Diagnosis of recurrent or refractory malignancy with histologic verification of malignancy at original diagnosis or relapse, except patients with extra-cranial germ-cell tumors who have elevations of serum tumor markers including alpha-fetoprotein or beta-HCG, and/or patients with intrinsic brain stem tumors or patients with CNS-germ cell tumors and elevations of CSF or serum tumor markers including alpha-fetoprotein or beta-HCG.
3. Have either measurable or evaluable disease. Evaluable disease is defined as an assessment of tumor that cannot be measured using a ruler or calipers, but can be used to determine disease progression or response (e.g., positive lesions on MIBG or bone scan, metastatic bone marrow disease, elevated tumor markers, or presence of a malignant pleural effusion)
4. Have current disease state for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life
5. Have Performance Level: Karnofsky ≥ 50% for patients >16 years of age and Lansky ≥50 for patients ≤16 years of age
6. Neurologic deficits in patients with CNS tumors must have been relatively stable for at least 7 days prior to study enrollment. Patients with CNS tumors who are receiving steroids must be on a stable or decreasing dose for at least 7 days prior to study entry. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
7. Have fully recovered from the acute clinically significant toxic effects of prior anti-cancer therapy

   * Myelosuppressive chemotherapy: On first day of treatment be at least 7 days after the last dose of myelosuppressive chemotherapy for single agent 9 ING 41, at least 21 days after the last dose of myelosuppressive chemotherapy for 9-ING-41 plus irinotecan
   * Hematopoietic growth factors: At least 14 days after the last dose of a long-acting growth factor or 7 days for short-acting growth factor
   * Biologic (anti-neoplastic agent): At least 7 days after the last dose of a biologic agent.
   * Monoclonal antibodies: At least 28 days after the last dose of a monoclonal antibody
   * At least 14 days after local palliative XRT (small port); At least 100 days must have elapsed if prior TBI, craniospinal XRT or if ≥ 50% radiation of pelvis; At least 42 days must have elapsed if other substantial BM radiation
   * Stem Cell Infusion without TBI: No evidence of active graft versus host disease and at least 84 days must have elapsed after transplant or stem cell infusion.
   * Patients undergoing a major surgical procedure or laparoscopic procedure are eligible for enrollment after at least 28 days of the procedure, 14 days after an open biopsy.
   * Patients undergoing a major surgical procedure, laparoscopic procedure or open biopsy are eligible for enrollment after at least 28 days of the procedure
   * Central line placement or subcutaneous port placement is not considered major surgery.
   * Core biopsy within 7 days prior to enrollment
   * Fine needle aspirate within 7 days prior to enrollment
   * Surgical or other wounds must be adequately healed prior to enrollment
8. Have received at least one front line treatment regimen for the treatment of their malignancy - on the Irinotecan combination arm, patients may have received prior Irinotecan
9. Have adequate organ and marrow function on first day of study treatment as follows:

   * For single agent 9-ING-41: ANC ≥ 500/mm3 For 9-ING-41 plus Irinotecan: ANC ≥ 1000/mm3
   * For single agent 9-ING-41: Platelets ≥ 50,000/mm3 For 9-ING-41 plus Irinotecan: Platelets ≥ 100,000/mm3
   * Hemoglobin ≥ 8 g/dL
   * Bilirubin ≤ 1.5 mg/dL
   * Alanine aminotransferase (ALT) ≤ 5.0 x upper limit of normal (ULN) unless elevation considered due to disease
   * Aspartate transaminase (AST) ≤ 5.0 x ULN unless elevation considered due to disease
   * Serum amylase and lipase ≤ 1.5 x ULN unless elevation considered due to disease
   * Creatinine clearance or radioisotope GFR ≥ 70 ml/min/1.73m2 or a serum creatinine based on age/gender as follows:

   Age Maximum Serum Creatinine (mg/dL) Maximum Serum Creatinine (mg/dL) Male Female 1 month to <6 months 0.4 0.4 6 months to <1 year 0.5 0.5 1 to <2 years 0.6 0.6 2 to <6 years 0.8 0.8 6 to <10 years 1 1 10 to <13 years 1.2 1.2 13 to <16 years 1.5 1.4

   ≥ 16 years 1.7 1.4
10. Pregnancy tests must be obtained in girls who are post-menarchal. Girls of childbearing potential must have a negative baseline blood or urine pregnancy test within 72 hours of first study therapy. Patients of childbearing potential must agree to use hormonal or barrier birth control with spermicidal gel, or total abstinence to avoid pregnancy for the duration of study participation and in the following 100 days after discontinuation of study treatment (see Section 4.1.1).
11. All patients and/or their parents or legal guardians must sign a written informed consent. The investigational nature and objectives of the trial, the procedures and treatments involved and their attendant risks and discomforts, and potential alternative therapies will be carefully explained to the patient or the patient's parents or guardian if the patient is a child, and a signed informed consent and assent will be obtained according to institutional guidelines

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from trial entry:

1. Has hypersensitivity to any of the components of 9-ING-41 and/or Irinotecan or to the excipients used in their formulation
2. Has uncontrolled concurrent illness that would limit compliance with study requirements
3. Has clinically significant retinal disease
4. Has current malignancy other than the target malignancy with the exception of surgically treated local tumors or is currently receiving other anti-cancer therapies, including radiation.
5. Has not recovered from clinically significant toxicities as a result of prior anticancer therapy, except alopecia, infertility and ototoxicity. Recovery is defined as ≤ Grade 2 severity per Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 (v5.0)
6. Is pregnant or lactating
7. Has received a prior solid organ transplantation
8. Is receiving any other investigational medicinal product or participating in another interventional clinical trial

Max Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5 | 3-12 months
  The standard assessments used to assign a score to any affected organ system as per the NCI CTCAE 5 will be conduced at each protocol-specified timepoint.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of California, San Francisco, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Chicago, Chicago, Illinois
  - Mott Children's Hospital, Ann Arbor, Michigan
  - Levine Cancer Center, Charlotte, North Carolina
  - Duke Children's Hospital and Health Center, Duke University Medical Center, Durham, North Carolina
  - Brown University, Providence, Rhode Island
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Research Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pal K, Cao Y, Gaisina IN, Bhattacharya S, Dutta SK, Wang E, Gunosewoyo H, Kozikowski AP, Billadeau DD, Mukhopadhyay D. Inhibition of GSK-3 induces differentiation and impaired glucose metabolism in renal cancer. Mol Cancer Ther. 2014 Feb;13(2):285-96. doi: 10.1158/1535-7163.MCT-13-0681. Epub 2013 Dec 10. PMID 24327518
- [Result] Ugolkov A, Gaisina I, Zhang JS, Billadeau DD, White K, Kozikowski A, Jain S, Cristofanilli M, Giles F, O'Halloran T, Cryns VL, Mazar AP. GSK-3 inhibition overcomes chemoresistance in human breast cancer. Cancer Lett. 2016 Oct 1;380(2):384-392. doi: 10.1016/j.canlet.2016.07.006. Epub 2016 Jul 14. PMID 27424289
- [Result] Ugolkov A, Qiang W, Bondarenko G, Procissi D, Gaisina I, James CD, Chandler J, Kozikowski A, Gunosewoyo H, O'Halloran T, Raizer J, Mazar AP. Combination Treatment with the GSK-3 Inhibitor 9-ING-41 and CCNU Cures Orthotopic Chemoresistant Glioblastoma in Patient-Derived Xenograft Models. Transl Oncol. 2017 Aug;10(4):669-678. doi: 10.1016/j.tranon.2017.06.003. Epub 2017 Jun 30. PMID 28672195
- [Result] Karmali R, Chukkapalli V, Gordon LI, Borgia JA, Ugolkov A, Mazar AP, Giles FJ. GSK-3beta inhibitor, 9-ING-41, reduces cell viability and halts proliferation of B-cell lymphoma cell lines as a single agent and in combination with novel agents. Oncotarget. 2017 Nov 11;8(70):114924-114934. doi: 10.18632/oncotarget.22414. eCollection 2017 Dec 29. PMID 29383130
- [Result] Ugolkov AV, Bondarenko GI, Dubrovskyi O, Berbegall AP, Navarro S, Noguera R, O'Halloran TV, Hendrix MJ, Giles FJ, Mazar AP. 9-ING-41, a small-molecule glycogen synthase kinase-3 inhibitor, is active in neuroblastoma. Anticancer Drugs. 2018 Sep;29(8):717-724. doi: 10.1097/CAD.0000000000000652. PMID 29846250
- [Result] Wu X, Stenson M, Abeykoon J, Nowakowski K, Zhang L, Lawson J, Wellik L, Li Y, Krull J, Wenzl K, Novak AJ, Ansell SM, Bishop GA, Billadeau DD, Peng KW, Giles F, Schmitt DM, Witzig TE. Targeting glycogen synthase kinase 3 for therapeutic benefit in lymphoma. Blood. 2019 Jul 25;134(4):363-373. doi: 10.1182/blood.2018874560. Epub 2019 May 17. PMID 31101621
- [Result] Ding L, Madamsetty VS, Kiers S, Alekhina O, Ugolkov A, Dube J, Zhang Y, Zhang JS, Wang E, Dutta SK, Schmitt DM, Giles FJ, Kozikowski AP, Mazar AP, Mukhopadhyay D, Billadeau DD. Glycogen Synthase Kinase-3 Inhibition Sensitizes Pancreatic Cancer Cells to Chemotherapy by Abrogating the TopBP1/ATR-Mediated DNA Damage Response. Clin Cancer Res. 2019 Nov 1;25(21):6452-6462. doi: 10.1158/1078-0432.CCR-19-0799. Epub 2019 Sep 18. PMID 31533931
- [Result] Jeffers A, Qin W, Owens S, Koenig KB, Komatsu S, Giles FJ, Schmitt DM, Idell S, Tucker TA. Glycogen Synthase Kinase-3beta Inhibition with 9-ING-41 Attenuates the Progression of Pulmonary Fibrosis. Sci Rep. 2019 Dec 12;9(1):18925. doi: 10.1038/s41598-019-55176-w. PMID 31831767
- [Result] Kuroki H, Anraku T, Kazama A, Bilim V, Tasaki M, Schmitt D, Mazar AP, Giles FJ, Ugolkov A, Tomita Y. 9-ING-41, a small molecule inhibitor of GSK-3beta, potentiates the effects of anticancer therapeutics in bladder cancer. Sci Rep. 2019 Dec 27;9(1):19977. doi: 10.1038/s41598-019-56461-4. PMID 31882719
- [Result] Walz A, Ugolkov A, Chandra S, Kozikowski A, Carneiro BA, O'Halloran TV, Giles FJ, Billadeau DD, Mazar AP. Molecular Pathways: Revisiting Glycogen Synthase Kinase-3beta as a Target for the Treatment of Cancer. Clin Cancer Res. 2017 Apr 15;23(8):1891-1897. doi: 10.1158/1078-0432.CCR-15-2240. Epub 2017 Jan 4. PMID 28053024